CLINICAL TRIAL: NCT02075047
Title: A PHASE 3, MULTICENTER, FOUR-WEEK, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP EFFICACY AND SAFETY TRIAL OF FLEXIBLE DOSES OF ORAL ZIPRASIDONE IN CHILDREN AND ADOLESCENTS WITH BIPOLAR I DISORDER (CURRENT OR MOST RECENT EPISODE MANIC)
Brief Title: Efficacy and Safety Trial of Flexible Doses of Oral Ziprasidone in Children and Adolescents With Bipolar I Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on recent input from FDA, the pre-specified final analysis will be performed at the current enrollment using a re-estimation of the sample size.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A1281198
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder (current or most recent episode manic). Children and adolescents aged 10 to 17 years.
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo oral capsules
- ziprasidone (Experimental)
  Interventions: Drug: ziprasidone oral capsules

INTERVENTIONS:
Drug: placebo oral capsules — Placebo matching the oral ziprasidone capsules of 20,40, 60 and 80 mg in strength. Subjects will be dosed for 4 weeks using a flexible dosing design. Dosing is stratified based on weight, with subjects <45 kg having a target dose range of 60-80 mg/day and subjects >/= 45 kg having a target dose range of 120-180 mg/day.
  Arms: 1
Drug: ziprasidone oral capsules — Oral ziprasidone capsules of 20,40, 60 and 80 mg in strength. Subjects will be dosed for 4 weeks using a flexible dosing design. Dosing is stratified based on weight, with subjects <45 kg having a target dose range of 60-80 mg/day and subjects >/= 45 kg having a target dose range of 120-180 mg/day.
  Arms: ziprasidone

SUMMARY:
The purpose of this study is to determine if ziprasidone is safe and effective for the treatment of children and adolescents (ages 10-17) with bipolar I disorder (manic or mixed).

ELIGIBILITY:
Inclusion Criteria:

* DSM V criteria for Bipolar I disorder (manic or mixed); age 10 - 17 years.

Exclusion Criteria:

* Imminent risk of suicide or homicide, as judged by the site investigator; any history of serious or unstable medical illness, including risk for QT prolongation.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2020-04-11 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (46):
  - Harmonex Neuroscience Research, Inc., Dothan, Alabama
  - Woodland International Research Group Inc., Little Rock, Arkansas
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - California Pharmaceutical Research Institute, Anaheim, California
  - NRC Research Institute, Orange, California
  - Asclepes Research Centers, Panorama City, California
  - University of California Davis Medical Center MIND Institute, Sacramento, California
  - Elite Clinical Trials, Incorporated, Wildomar, California
  - Children's National Health System, Washington D.C., District of Columbia
  - Da Vinci Research Institute Inc, Boca Raton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - APG Research LLC, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Inova Clinical Trials and Research Centre, Fayetteville, Georgia
  - Attalla Consultants, LLC dba Institute for Behavioral Medicine, Smyrna, Georgia
  - Sleep and Behavior Medicine Institute, Vernon Hills, Illinois
  - Hugo W. Moser Research Institute at Kennedy Krieger Institute Clinical Trials Unit, Baltimore, Maryland
  - Kennedy Krieger Institute Inpatient Clinic, Baltimore, Maryland
  - Kennedy Krieger Institute Outpatient Clinic, Baltimore, Maryland
  - Psychiatric Mental Health Program at Kennedy Krieger Institute Clinical Trials Unit, Baltimore, Maryland
  - Johns Hopkins Hospital Pediatric Clinical Research Unit, Baltimore, Maryland
  - Charlotte R. Bloomberg Children's Center, Baltimore, Maryland
  - Johns Hopkins Hospital Investigational Drug Services, Baltimore, Maryland
  - Clinical Research Integrity(CRI) Lifetree, LLC, Marlton, New Jersey
  - Erie County Medical Center/State University of New York (SUNY) at Buffalo Affiliate, Buffalo, New York
  - The Zucker Hillside Hospital Northwell Health, Glen Oaks, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - UT Health Science Center at Houston (UTHSC-H), Houston, Texas
  - AIM Trials, Plano, Texas
  - Research Across America, Plano, Texas
  - Family Psychiatry Of The Woodlands, The Woodlands, Texas
  - Fontaine Medical Laboratories, Charlottesville, Virginia
  - Northridge Medical Plaza, Charlottesville, Virginia
  - University of Virginia Center for Psychopharmacology Research in Youth, Charlottesville, Virginia
  - UVA Child & Family Psychiatry Clinic, Charlottesville, Virginia
  - Clinical Research Partners, LLC, Petersburg, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Eastside Therapeutic Resource dba Core Clinical Research, Everett, Washington
- Ukraine (4):
  - Communal Non profit Enterprise "City Children Clinical Hospital #5 of Dnipro Regional Council", Dnipro
  - Communal Nonprofit Enterprise "City Children Clinical Hospital #5 of Dnipro Regional Council, Dnipro
  - Communal Nonprofit Enterprise "Odesa Regional Medical Centre of Mental Health" of Odesa, Odesa
  - Municipal Institution "Vinnytsya Regional Psychoneurologycal Hospital Named After O.I. Yushenko", Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Findling RL, Atkinson S, Bachinsky M, Raiter Y, Abreu P, Ianos C, Chappell P. Efficacy, Safety, and Tolerability of Flexibly Dosed Ziprasidone in Children and Adolescents with Mania in Bipolar I Disorder: A Randomized Placebo-Controlled Replication Study. J Child Adolesc Psychopharmacol. 2022 Apr;32(3):143-152. doi: 10.1089/cap.2021.0121. Epub 2022 Apr 7. PMID 35394365
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281198&StudyName=Efficacy%20and%20Safety%20Trial%20of%20Flexible%20Doses%20of%20Oral%20Ziprasidone%20in%20Children%20and%20Adolescents%20with%20Bipolar%20I%20Disorder%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in the United States and Ukraine. Study started on 23 May 2014 and completed on 18 May 2020. Total 171 participants were randomized to treatment, of which 86 received study medication.
Groups:
- Ziprasidone: Participants were randomized to receive ziprasidone capsules orally once daily for 4 weeks. Dose was titrated over the first 7-14 days of treatment, and the stable dose was maintained for remaining treatment period. Participants with body weight less than 45 kilogram (kg) received 60 to 80 milligram per day (mg/day) and participants with body weight greater than or equal to (>=) 45 kg received 120 to 160 mg/day, as per investigator discretion. Participants after completion or discontinuation of treatment were followed-up to 35 days (5 weeks) after last dose in this study or were eligible to enroll in open label extension study A1281201 (NCT03768726).
- Placebo: Participants were randomized to receive placebo capsules matched to ziprasidone once daily for 4 weeks. Participants after completion or discontinuation of treatment were followed-up to 35 days (5 weeks) after last dose in this study or were eligible to enroll in open label extension study A1281201 (NCT03768726).
Period: Treatment Phase (4 Weeks)
Arm/Group | Ziprasidone | Placebo
Started | 86 | 85
Completed | 63 | 75
Not Completed | 23 | 10
Not completed — Adverse Event | 14 | 4
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Medication Error Without Associated Adverse Event | 1 | 0
Not completed — Screen Failure | 1 | 0
Not completed — Other | 1 | 1
Not completed — Withdrawal By Parent/Guardian | 4 | 2
Period: Follow up Phase (5 Weeks)
Arm/Group | Ziprasidone | Placebo
Started | 86 (Participants were followed up after completion or discontinuation of treatment.) | 85 (Participants were followed up after completion or discontinuation of treatment.)
Completed | 60 | 72
Not Completed | 26 | 13
Not completed — Adverse Event | 14 | 4
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Medication Error Without Associated Adverse Event | 1 | 0
Not completed — Screen Failure | 1 | 0
Not completed — Other | 1 | 2
Not completed — Withdrawal By Parent/Guardian | 7 | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and took at least 1 dose of study medication (ziprasidone or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Customized [Count of Participants; unit: Participants]
  10 - >14 Years | 46 | 44 | 90
  14-17 Years | 40 | 41 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 95
  Male | 38 | 38 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 26
  Not Hispanic or Latino | 74 | 71 | 145
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 59 | 55 | 114
  Race: Black or African American | 23 | 24 | 47
  Race: Asian | 1 | 1 | 2
  Race: Other | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score at Week 4
Description: YMRS: an 11-item scale that measured the severity of manic episodes. Four items (irritability, speech, thought content, and disruptive/ aggressive behavior) were rated on a scale from 0 (symptom absent) to 8 (symptom extremely severe). The remaining items were rated on a scale from 0 (symptom absent) to 4 (symptom extremely severe). YMRS total score was sum of score of all 11 items and ranged from 0 (no symptoms) to 60 (extreme severity of symptoms), higher score indicated higher severity of mania.
Time Frame: Baseline, Week 4
Population: Intent-to-treat (ITT) included all randomized participants who had baseline measurements, took at least 1 dose of study medication (ziprasidone or placebo) and had at least 1 post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
units on a scale | -16.51 (1.15) | -12.29 (1.10)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Change at Week 4: Results were obtained from a mixed effects repeated measures analysis of covariance model treatment, visit, visit-by-treatment interaction, and weight category as fixed effects and baseline score as a covariate along with participant as a random effect; Test type: Superiority; p = 0.005, Mixed Models Analysis; Difference in least square (LS) mean = -4.23, 95% CI 2-sided [-7.14 to -1.32], Standard Error of Mean 1.47

2. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at Weeks 1, 2, 3, and 4
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill), higher scores indicated more severity of illness.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: ITT included all randomized participants who had baseline measurements, took at least 1 dose of study medication (ziprasidone or placebo) and had at least 1 post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
units on a scale
  Change at Week 1 | -0.91 (0.10) | -0.47 (0.10)
  Change at Week 2 | -1.13 (0.12) | -0.91 (0.12)
  Change at Week 3 | -1.53 (0.13) | -1.14 (0.13)
  Change at Week 4 | -1.59 (0.14) | -1.32 (0.14)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Change at Week 1: Results were obtained from a mixed effects repeated measures analysis of covariance model treatment, visit, visit-by-treatment interaction, and weight category as fixed effects and baseline score as a covariate along with participant as a random effect; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in LS mean = -0.45, 95% CI 2-sided [-0.69 to -0.20], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Change at Week 2: Results were obtained from a mixed effects repeated measures analysis of covariance model treatment, visit, visit-by-treatment interaction, and weight category as fixed effects and baseline score as a covariate along with participant as a random effect; Test type: Superiority; p = 0.174, Mixed Models Analysis; Difference in LS mean = -0.22, 95% CI 2-sided [-0.53 to 0.10], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Change at Week 3: Results were obtained from a mixed effects repeated measures analysis of covariance model treatment, visit, visit-by-treatment interaction, and weight category as fixed effects and baseline score as a covariate along with participant as a random effect; Test type: Superiority; p = 0.024, Mixed Models Analysis; Difference in LS mean = -0.38, 95% CI 2-sided [-0.71 to -0.05], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.138, Mixed Models Analysis; Difference in LS mean = -0.28, 95% CI 2-sided [-0.64 to 0.09], Standard Error of Mean 0.19

3. Secondary Outcome: Change From Baseline in the Young Mania Rating Scale (YMRS) Total Score at Weeks 1, 2, and 3
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
units on a scale
  Change at Week 1 | -11.43 (0.94) | -5.58 (0.93)
  Change at Week 2 | -13.70 (1.02) | -9.53 (1.01)
  Change at Week 3 | -16.79 (1.04) | -11.17 (1.01)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in LS mean = -5.85, 95% CI 2-sided [-8.16 to -3.54], Standard Error of Mean 1.17
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.002, Mixed Models Analysis; Difference in LS mean = -4.17, 95% CI 2-sided [-6.74 to -1.59], Standard Error of Mean 1.30
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in LS mean = -5.63, 95% CI 2-sided [-8.21 to -3.04], Standard Error of Mean 1.31

4. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Scores at Weeks 1, 2, 3, and 4
Description: CGI-I: 7-point clinician rated scale which rates the participant's improvement or worsening from baseline, ranging from 1 (very much improved) to 7 (very much worse), higher scores indicate less improvement.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
units on a scale
  Change at Week 1 | 2.89 (0.11) | 3.41 (0.11)
  Change at Week 2 | 2.75 (0.12) | 2.89 (0.12)
  Change at Week 3 | 2.42 (0.12) | 2.68 (0.12)
  Change at Week 4 | 2.30 (0.13) | 2.64 (0.13)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Change at Week 1: Results were obtained from a mixed effects repeated measures analysis of covariance model treatment, visit, visit-by-treatment interaction, and weight category as fixed effects along with participant as a random effect; Test type: Superiority; p = 0.001, Mixed Models Analysis; Difference in LS mean = -0.52, 95% CI 2-sided [-0.78 to -0.26], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Change at Week 2: Results were obtained from a mixed effects repeated measures analysis of covariance model treatment, visit, visit-by-treatment interaction, and weight category as fixed effects along with participant as a random effect; Test type: Superiority; p = 0.349, Mixed Models Analysis; Difference in LS mean = -0.15, 95% CI 2-sided [-0.45 to 0.16], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Change at Week 3: Results were obtained from a mixed effects repeated measures analysis of covariance model treatment, visit, visit-by-treatment interaction, and weight category as fixed effects along with participant as a random effect; Test type: Superiority; p = 0.103, Mixed Models Analysis; Difference in LS mean = -0.26, 95% CI 2-sided [-0.57 to 0.05], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; Change at Week 4: Results were obtained from a mixed effects repeated measures analysis of covariance model treatment, visit, visit-by-treatment interaction, and weight category as fixed effects along with participant as a random effect; Test type: Superiority; p = 0.044, Mixed Models Analysis; Difference in LS mean = -0.35, 95% CI 2-sided [-0.68 to -0.01], Standard Error of Mean 0.17

5. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/ incapacity; congenital anomaly. AEs included both serious and all non-serious AEs.
Time Frame: Screening (2 Weeks prior to Day 1) up to maximum of 5 Weeks after administration of the final dose of study medication (maximum up to 11 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
Participants
  AEs | 67 | 50
  SAEs | 3 | 0

6. Other Pre Specified Outcome: Number of Participants With Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categorization Mapped From Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS: a measure used to identify and assess participants at risk for suicide. It is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors. C-SSRS items were mapped to the following C-CASA categories: completed suicide, attempted suicide (actual attempt; aborted attempt; interrupted attempt), non-suicidal self-injurious behavior, preparatory acts, suicidal ideation (wish to be dead; non-specific active suicidal thoughts; active suicidal ideation with any methods [not plan], without intent to act; active suicidal ideation with some intent to act, without specific plan; active suicidal ideation with specific plan and intent; self-injurious behavior, no suicidal intent). Rows according to C-CASA categories at specified time points are reported in this outcome measure, only when there was non-zero data/values for at least 1 reporting arm.
Time Frame: Screening (2 Weeks prior to Day 1), Baseline (Day 1), Week 1, 2, 3, 4, Early Termination Visit (anytime from Day 1 to Week 4), Follow up Visit (anytime from Day 1 up to 5 weeks after last dose of study drug = anytime from Day 1 to Week 9)
Population: ITT included all randomized participants who had baseline measurements, took at least 1 dose of study medication (ziprasidone or placebo) and had at least 1 post-baseline visit. Here 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
Participants
  Screening: Actual Attempt | 5 | 3
  Screening: Interrupted Attempt | 0 | 1
  Screening: Non-Suicidal Self-Injurious Behavior | 10 | 5
  Screening: Preparatory Acts | 0 | 1
  Screening: Wish To Be Dead | 25 | 25
  Screening: Non-specific Active Suicidal Thoughts | 16 | 13
  Baseline: Wish To Be Dead | 1 | 0
  Baseline: Active Suicidal Thoughts With No Plan, Intent | 4 | 7
  Baseline: Active Suicidal Thoughts With No Plan, Some Intent | 2 | 3
  Baseline: Active Suicidal Thoughts With Plan, Intent | 4 | 3
  Week 1: Wish To Be Dead: number analyzed (Participants) | 78 | 83
  Week 1: Wish To Be Dead | 0 | 1
  Week 4: Non-Suicidal Self-Injurious Behavior: number analyzed (Participants) | 63 | 75
  Week 4: Non-Suicidal Self-Injurious Behavior | 1 | 0
  Week 4: Wish To Be Dead: number analyzed (Participants) | 63 | 75
  Week 4: Wish To Be Dead | 2 | 0
  Week 4: Non-specific Active Suicidal Thoughts: number analyzed (Participants) | 63 | 75
  Week 4: Non-specific Active Suicidal Thoughts | 1 | 0
  Early Termination: Wish To Be Dead: number analyzed (Participants) | 21 | 5
  Early Termination: Wish To Be Dead | 1 | 0
  Early Termination: Non-specific Active Suicidal Thoughts: number analyzed (Participants) | 21 | 5
  Early Termination: Non-specific Active Suicidal Thoughts | 1 | 0
  Early Termination: Active Suicidal Thoughts With No Plan, Intent: number analyzed (Participants) | 21 | 5
  Early Termination: Active Suicidal Thoughts With No Plan, Intent | 1 | 0
  Follow up: Actual Attempt: number analyzed (Participants) | 62 | 64
  Follow up: Actual Attempt | 1 | 0
  Follow up: Wish To Be Dead: number analyzed (Participants) | 62 | 64
  Follow up: Wish To Be Dead | 2 | 0

7. Other Pre Specified Outcome: Number of Participants Who Took at Least 1 Concomitant Medication and Concomitant Non-Drug Treatments/Procedures
Description: Concomitant medications or treatments were those prescription and over-the-counter drugs and supplements or non drug treatment/procedures other than the study medication.
Time Frame: Screening (2 Weeks prior to Day 1) up to 1 Week after administration of the final dose of study medication (maximum for 7 Weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
Participants
  Concomitant Medication | 55 | 47
  Concomitant Non-Drug Treatments/Procedures | 6 | 7

8. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria: Hematology-hemoglobin(Hg),hematocrit,erythrocytes(ery)<0.8*LLN,ery mean corpuscular volume <0.9*LLN>1.1*ULN,platelets<0.5*LLN>1.75*ULN,leukocytes(leu)<0.6*LLN>1.5*ULN,lymphocytes(lym),lym/leu,neutrophils(neu),neu/leu<0.8*LLN>1.2*ULN,basophils (bas),bas/leu, eosinophils(eos), eos/leu, monocytes(mon),mon/leu>1.2*ULN; Clinical chemistry bilirubin: total, direct, indirect>1.5*ULN, aspartate aminotransferase,alanine aminotransferase, gamma glutamyl transferase, lactate dehydrogenase,alkaline phosphatase>3.0*ULN,protein,albumin<0.8*LLN>1.2*ULN,blood urea nitrogen,creatinine>1.3*ULN, urate>1.2*ULN,HDL<0.8*LLN;LDL>1.2*ULN cholesterol(CH),sodium<0.95*LLN>1.05*ULN,potassium, chloride,calcium,magnesium,bicarbonate<0.9*LLLN>1.1*ULN,phosphate,free thyroxine,thyroid stimulating hormone<0.8*LLN>1.2*ULN,prolactin>1.1*ULN,glucose<0.6*LLN>1.5*ULN,HgA1C,CH, triglycerides>1.3*ULN,creatine kinase>2.0*ULN; Urinalysis-specific gravity<1.003>1.030,pH<4.5 >8,urine glucose, protein, Hg, ketones:>=1.
Time Frame: as for outcome 7
Population: The safety analysis set included all participants who were randomized and took at least 1 dose of study medication (ziprasidone or placebo). Here 'Overall Number of Participants Analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 84 | 83
Participants | 50 | 62

9. Other Pre Specified Outcome: Number of Participants With Physical Examination Abnormalities
Description: Parameters assessed for physical examination included: oral/tympanic temperature, general appearance, skin, head, ears, eyes, nose, throat, heart, lungs, breasts (if medically indicated), abdomen, external genitalia [if medically indicated], extremities, back/spinal system, lymph nodes or worsening of medical history conditions. Abnormality in physical examination was at the investigator's discretion.
Time Frame: Screening (2 Weeks prior to Day 1) up to Week 4
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
Participants | 4 | 5

10. Other Pre Specified Outcome: Change From Baseline in Blood Pressure at Week 1, 2, 3, 4, Early Termination Visit and Follow-up Visit
Description: Change from baseline in sitting and standing systolic blood pressure and diastolic blood pressure in millimeter of mercury (mmHg) was reported.
Time Frame: Baseline, Week 1, 2, 3, 4, Early Termination Visit (anytime from Day 1 to Week 4), Follow up Visit (anytime from Day 1 up to 5 weeks after last dose of study drug = anytime from Day 1 to Week 9)
Population: The safety analysis set included all participants who were randomized and took at least 1 dose of study medication (ziprasidone or placebo). Here 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
millimeter of mercury
  Sitting Systolic Blood Pressure, Baseline | 110.5 (9.84) | 110.9 (11.45)
  Sitting Systolic Blood Pressure, Change at Week 1: number analyzed (Participants) | 78 | 83
  Sitting Systolic Blood Pressure, Change at Week 1 | 0.7 (6.90) | 0.2 (8.71)
  Sitting Systolic Blood Pressure, Change at Week 2: number analyzed (Participants) | 67 | 78
  Sitting Systolic Blood Pressure, Change at Week 2 | 0.2 (9.65) | 0.1 (9.26)
  Sitting Systolic Blood Pressure, Change at Week 3: number analyzed (Participants) | 64 | 75
  Sitting Systolic Blood Pressure, Change at Week 3 | -0.7 (10.12) | -0.6 (8.93)
  Sitting Systolic Blood Pressure, Change at Week 4: number analyzed (Participants) | 63 | 75
  Sitting Systolic Blood Pressure, Change at Week 4 | -0.7 (10.60) | -2.2 (10.39)
  Sitting Systolic Blood Pressure, Change at Early Termination: number analyzed (Participants) | 20 | 5
  Sitting Systolic Blood Pressure, Change at Early Termination | 0.7 (7.87) | 6.4 (5.90)
  Sitting Systolic Blood Pressure, Change at Follow up: number analyzed (Participants) | 21 | 22
  Sitting Systolic Blood Pressure, Change at Follow up | -1.4 (12.44) | -2.2 (8.35)
  Standing Systolic Blood Pressure, Baseline | 110.7 (9.53) | 112.0 (10.16)
  Standing Systolic Blood Pressure, Change at Week 1: number analyzed (Participants) | 78 | 83
  Standing Systolic Blood Pressure, Change at Week 1 | 0.8 (7.67) | -2.5 (10.38)
  Standing Systolic Blood Pressure, Change at Week 2: number analyzed (Participants) | 67 | 78
  Standing Systolic Blood Pressure, Change at Week 2 | 0.1 (9.13) | -1.8 (9.71)
  Standing Systolic Blood Pressure, Change at Week 3: number analyzed (Participants) | 64 | 75
  Standing Systolic Blood Pressure, Change at Week 3 | -0.1 (9.68) | -1.8 (9.71)
  Standing Systolic Blood Pressure, Change at Week 4: number analyzed (Participants) | 63 | 75
  Standing Systolic Blood Pressure, Change at Week 4 | -0.8 (9.50) | -2.5 (10.77)
  Standing Systolic Blood Pressure, Change at Early Termination: number analyzed (Participants) | 20 | 5
  Standing Systolic Blood Pressure, Change at Early Termination | -2.1 (10.14) | 5.6 (13.58)
  Standing Systolic Blood Pressure, Change at Follow up: number analyzed (Participants) | 21 | 22
  Standing Systolic Blood Pressure, Change at Follow up | -4.9 (11.86) | -4.4 (10.01)
  Sitting Diastolic Blood Pressure, Baseline | 68.8 (7.99) | 70.3 (7.94)
  Sitting Diastolic Blood Pressure, Change at Week 1: number analyzed (Participants) | 78 | 83
  Sitting Diastolic Blood Pressure, Change at Week 1 | 0.7 (7.72) | -1.5 (8.49)
  Sitting Diastolic Blood Pressure, Change at Week 2: number analyzed (Participants) | 67 | 78
  Sitting Diastolic Blood Pressure, Change at Week 2 | 1.0 (9.76) | -0.6 (9.40)
  Sitting Diastolic Blood Pressure, Change at Week 3: number analyzed (Participants) | 64 | 75
  Sitting Diastolic Blood Pressure, Change at Week 3 | 0.2 (9.36) | 0.1 (8.03)
  Sitting Diastolic Blood Pressure, Change at Week 4: number analyzed (Participants) | 63 | 75
  Sitting Diastolic Blood Pressure, Change at Week 4 | 1.1 (8.18) | -0.6 (10.22)
  Sitting Diastolic Blood Pressure, Change at Early Termination: number analyzed (Participants) | 20 | 5
  Sitting Diastolic Blood Pressure, Change at Early Termination | -1.8 (9.65) | 2.0 (8.46)
  Sitting Diastolic Blood Pressure, Change at Follow up: number analyzed (Participants) | 21 | 22
  Sitting Diastolic Blood Pressure, Change at Follow up | 2.7 (8.64) | 1.7 (6.75)
  Standing Diastolic Blood Pressure, Baseline | 70.3 (6.98) | 72.3 (7.91)
  Standing Diastolic Blood Pressure, Change at Week 1: number analyzed (Participants) | 78 | 83
  Standing Diastolic Blood Pressure, Change at Week 1 | 1.5 (7.40) | -1.6 (8.46)
  Standing Diastolic Blood Pressure, Change at Week 2: number analyzed (Participants) | 67 | 78
  Standing Diastolic Blood Pressure, Change at Week 2 | -0.1 (7.83) | -1.7 (8.75)
  Standing Diastolic Blood Pressure, Change at Week 3: number analyzed (Participants) | 64 | 75
  Standing Diastolic Blood Pressure, Change at Week 3 | -1.1 (7.91) | -1.6 (10.27)
  Standing Diastolic Blood Pressure, Change at Week 4: number analyzed (Participants) | 63 | 75
  Standing Diastolic Blood Pressure, Change at Week 4 | 1.0 (7.76) | -0.5 (9.83)
  Standing Diastolic Blood Pressure, Change at Early Termination: number analyzed (Participants) | 20 | 5
  Standing Diastolic Blood Pressure, Change at Early Termination | 1.3 (10.22) | 1.6 (7.60)
  Standing Diastolic Blood Pressure, Change at Follow up: number analyzed (Participants) | 21 | 22
  Standing Diastolic Blood Pressure, Change at Follow up | 1.2 (8.41) | -2.1 (12.89)

11. Other Pre Specified Outcome: Change From Baseline in Pulse Rate at Week 1, 2, 3, 4, Early Termination Visit and Follow-up Visit
Description: Change from baseline pulse rate in (beats per minute) was reported in sitting and standing positions.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
beats per minute
  Sitting, Baseline | 79.1 (12.58) | 75.8 (9.80)
  Sitting, Change at Week 1: number analyzed (Participants) | 78 | 83
  Sitting, Change at Week 1 | -0.9 (11.24) | -2.0 (9.40)
  Sitting, Change at Week 2: number analyzed (Participants) | 67 | 78
  Sitting, Change at Week 2 | -2.4 (11.75) | 1.5 (8.82)
  Sitting, Change at Week 3: number analyzed (Participants) | 64 | 75
  Sitting, Change at Week 3 | -0.5 (12.79) | 2.3 (10.61)
  Sitting, Change at Week 4: number analyzed (Participants) | 63 | 75
  Sitting, Change at Week 4 | -2.3 (11.49) | -0.2 (10.30)
  Early Termination: Sitting: number analyzed (Participants) | 20 | 5
  Early Termination: Sitting | 3.5 (14.02) | 1.6 (7.02)
  Follow up: Sitting: number analyzed (Participants) | 21 | 22
  Follow up: Sitting | 2.0 (11.32) | 3.1 (11.73)
  Standing, Baseline | 84.6 (12.23) | 83.3 (10.95)
  Standing, Change at Week 1: number analyzed (Participants) | 78 | 83
  Standing, Change at Week 1 | 2.1 (10.77) | -2.2 (10.18)
  Standing, Change at Week 2: number analyzed (Participants) | 67 | 78
  Standing, Change at Week 2 | -0.4 (12.25) | 1.9 (10.19)
  Standing, Change at Week 3: number analyzed (Participants) | 64 | 75
  Standing, Change at Week 3 | 1.4 (13.54) | 2.6 (11.70)
  Standing, Change at Week 4: number analyzed (Participants) | 63 | 75
  Standing, Change at Week 4 | -0.7 (11.77) | -0.6 (12.83)
  Early Termination: Standing: number analyzed (Participants) | 20 | 5
  Early Termination: Standing | 7.9 (13.98) | -6.2 (21.12)
  Follow up: Standing: number analyzed (Participants) | 21 | 22
  Follow up: Standing | 5.4 (10.15) | 4.5 (11.67)

12. Other Pre Specified Outcome: Change From Baseline in Height and Waist Circumference at Week 4 and Early Termination Visit
Description: Change from baseline in height and waist circumference in centimeter (cm) was reported.
Time Frame: Baseline, Week 4, Early Termination Visit (anytime from Day 1 to Week 4)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
centimeter
  Height, Baseline | 157.9 (10.63) | 159.7 (11.41)
  Height, Change at Week 4: number analyzed (Participants) | 63 | 75
  Height, Change at Week 4 | 0.4 (0.60) | 0.7 (1.77)
  Height, Change at Early Termination: number analyzed (Participants) | 19 | 5
  Height, Change at Early Termination | 0.2 (0.54) | 0.5 (0.73)
  Waist Circumference, Baseline | 76.9 (12.22) | 74.9 (10.56)
  Waist Circumference, Change at Week 4: number analyzed (Participants) | 63 | 75
  Waist Circumference, Change at Week 4 | -0.1 (2.79) | 0.3 (3.26)
  Waist Circumference, Change at Early Termination: number analyzed (Participants) | 19 | 5
  Waist Circumference, Change at Early Termination | 0.4 (3.77) | 1.0 (1.74)

13. Other Pre Specified Outcome: Change From Baseline in Body Weight at Week 4 and Early Termination Visit
Description: Change from baseline in body weight in kilogram (kg) was reported.
Time Frame: Baseline, Week 4, Early Termination Visit (anytime from Day 1 to Week 4)
Population: The safety analysis set included all participants who were randomized and took at least 1 dose of study medication (ziprasidone or placebo). Here 'number analyzed' signifies number of participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
kilogram
  Baseline | 57.5 (14.52) | 58.0 (14.54)
  Change at Week 4: number analyzed (Participants) | 63 | 75
  Change at Week 4 | 0.3 (1.97) | 0.8 (2.04)
  Change at Early Termination: number analyzed (Participants) | 19 | 5
  Change at Early Termination | -0.3 (1.75) | 1.0 (1.46)

14. Other Pre Specified Outcome: Change From Baseline in Body Mass Index (BMI) at Week 4 and Early Termination Visit
Description: Change from baseline in BMI in kilogram per meter square (kg/m^2) was reported.
Time Frame: Baseline, Week 4, Early Termination Visit (anytime from Day 1 to Week 4)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: kilogram per meter square
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
kilogram per meter square
  Baseline | 22.8 (4.15) | 22.5 (3.76)
  Change at Week 4: number analyzed (Participants) | 63 | 75
  Change at Week 4 | 0.1 (0.79) | 0.2 (0.92)
  Change at Early Termination: number analyzed (Participants) | 19 | 5
  Change at Early Termination | -0.3 (0.95) | 0.3 (0.51)

15. Other Pre Specified Outcome: Change From Baseline in Body Mass Index (BMI) Z-score at Week 4 and Early Termination Visit
Description: BMI z-score was reported using the Children's Hospital of Philadelphia z-score calculator. Z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher BMI.
Time Frame: Baseline, Week 4, Early Termination Visit (anytime from Day 1 to Week 4)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 86 | 85
z-score
  Baseline | 0.8 (0.87) | 0.7 (0.82)
  Change at Week 4: number analyzed (Participants) | 63 | 75
  Change at Week 4 | 0.0 (0.18) | -0.0 (0.24)
  Change at Early Termination: number analyzed (Participants) | 19 | 5
  Change at Early Termination | -0.0 (0.15) | -0.0 (0.22)

16. Other Pre Specified Outcome: Number of Participants With Pre-defined Categories of Electrocardiogram (ECG) Findings
Description: Pre-defined categories for ECG were: heart rate intervals - QT interval corrected using the Fridericia's formula (QTCF) value greater than or equal to (>=450) millisecond (msec), >=460 msec, >=480 msec, >=500 msec, >=30 msec increase, >=60 msec increase, >=75 msec increase, QT interval corrected using the Bazett's correction (QTCB) value >=450 msec, >=460 msec, >=480 msec, >=500 msec, >=30 msec increase, >=60 msec increase, >=75 msec increase, PR value >=25 percentage increase, QRS value >=25 percentage increase, QT value >=25 percentage increase, Respiratory rate (RR) value >=25 percentage increase, and Heart rate (HR) value >=25 percentage increase. Rows according to ECG pre-defined categories are reported in this outcome measure, only when there was non-zero data/values for at least 1 reporting arm.
Time Frame: as for outcome 7
Population: The safety analysis set included all participants who were randomized and took at least 1 dose of study medication (ziprasidone or placebo). Here ' Overall Number of Participants Analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
Participants
  QTcF at >=450 msec | 3 | 1
  QTcF at >=460 msec | 1 | 0
  QTcF at >=30 msec increase | 9 | 4
  QTcB at >=450 msec | 14 | 7
  QTcB at >=460 msec | 8 | 3
  QTcB at >=480 msec | 1 | 0
  QTcB at >=30 msec increase | 16 | 7
  QRS at >=25% increase | 3 | 1
  RR at >=25% increase | 12 | 14
  HR at >=25% increase | 18 | 9

17. Other Pre Specified Outcome: Change From Baseline in Children's Depression Rating Scale (CDRS-R) Total Score at Weeks 1, 2, 3, and 4 and Early Termination Visit
Description: CDRS-R: clinician-rated interview-based scale (with both child and parent or guardian) to assess 17 distinct symptom areas to derive an index of depression severity. Discrepancies between informants responses were resolved by using most impaired rating given by valid informant. Rated on a 7-point scale; range from 1 (no impairment) to 7 (maximum impairment). Higher scores indicated greater impairment. Total score calculated as sum of the 17 items ranged from 17 (no impairment) to 119 (maximum impairment); higher score indicated greater impairment.
Time Frame: Baseline, Week 1, 2, 3, 4, Early Termination Visit (anytime from Day 1 to Week 4)
Population: ITT included all randomized participants who had baseline measurements, took at least 1 dose of study medication (ziprasidone or placebo) and had at least 1 post-baseline visit. Here 'number analyzed' signifies number of participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
units on a scale
  Baseline | 29.0 (6.62) | 28.3 (5.74)
  Change at Week 1: number analyzed (Participants) | 78 | 83
  Change at Week 1 | -2.5 (5.78) | -0.8 (4.85)
  Change at Week 2: number analyzed (Participants) | 67 | 78
  Change at Week 2 | -2.9 (6.31) | -2.4 (5.37)
  Change at Week 3: number analyzed (Participants) | 64 | 75
  Change at Week 3 | -3.7 (6.39) | -3.3 (6.15)
  Change at Week 4: number analyzed (Participants) | 63 | 75
  Change at Week 4 | -3.6 (6.53) | -3.8 (5.99)
  Change at Early Termination: number analyzed (Participants) | 20 | 5
  Change at Early Termination | 2.3 (10.46) | -1.2 (4.60)

18. Other Pre Specified Outcome: Change From Baseline in Simpson-Angus Rating Scale (SARS) Total Score at Weeks 1, 2, 3, and 4
Description: SARS: 10-item clinician rated instrument to assess parkinsonian symptoms and related extrapyramidal side effects. All 10 items were anchored on a 5-point scale: range 0 (absence of condition, normal) to 4 (the most extreme form of condition). Total SARS score is sum of all individual item scores, and ranged from 0 (normal) to 40 (most extreme symptoms and effects); higher score indicates more affected.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
units on a scale
  Change at Week 1 | 0.09 (0.04) | -0.01 (0.04)
  Change at Week 2 | 0.11 (0.05) | -0.00 (0.05)
  Change at Week 3 | 0.11 (0.05) | -0.00 (0.05)
  Change at Week 4 | 0.09 (0.04) | -0.00 (0.04)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.050, Mixed Models Analysis; Difference in LS mean = 0.10, 95% CI 2-sided [0.00 to 0.20], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.124, Mixed Models Analysis; Difference in LS mean = 0.11, 95% CI 2-sided [-0.03 to 0.25], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.084, Mixed Models Analysis; Difference in LS mean = 0.11, 95% CI 2-sided [-0.01 to 0.23], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.104, Mixed Models Analysis; Difference in LS mean = 0.09, 95% CI 2-sided [-0.02 to 0.20], Standard Error of Mean 0.05

19. Other Pre Specified Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BAS): Global Clinical Assessment of Akathisia Subscale Score at Weeks 1, 2, 3, and 4
Description: BAS: clinician rated scale to assess akathisia by determining the degree of subjective restlessness and distress associated with restlessness. First 3 items (objective, subjective, and distress related to restlessness) were rated on a 4-point scale with range 0 (no symptoms) to 3 (maximum severity of symptoms). Item 4, global clinical assessment of akathisia subscale, was rated on a 6-point scale, and ranged from 0 (no symptoms) to 5 (maximum severity of symptoms); higher score indicates increased severity.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
units on a scale
  Change at Week 1 | -0.01 (0.01) | 0.02 (0.01)
  Change at Week 2 | 0.04 (0.03) | 0.04 (0.03)
  Change at Week 3 | 0.01 (0.02) | 0.01 (0.01)
  Change at Week 4 | 0.01 (0.01) | -0.01 (0.01)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.169, Mixed Models Analysis; Difference in LS mean = -0.02, 95% CI 2-sided [-0.06 to 0.01], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.893, Mixed Models Analysis; Difference in LS mean = -0.01, 95% CI 2-sided [-0.10 to 0.08], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.915, Mixed Models Analysis; Difference in LS mean = 0.00, 95% CI 2-sided [-0.04 to 0.04], Standard Error of Mean 0.02
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.289, Mixed Models Analysis; Difference in LS mean = 0.02, 95% CI 2-sided [-0.01 to 0.04], Standard Error of Mean 0.01

20. Other Pre Specified Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) - Movement Cluster Score at Weeks 1, 2, 3, and 4
Description: AIMS: clinician rated 12-item scale to document occurrences of dyskinesia in participants, specifically tardive dyskinesia. Items 1 to 10, scored as 0 (none) to 4 (severe); higher score indicates greater severity. Items 11 to 12 are questions with No or Yes response. Only the sum of the first 7 items were calculated to evaluate AIMS movement cluster score, giving a score range of 0 (none) to 28 (maximum severity), higher score indicates greater severity.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 85 | 83
units on a scale
  Change at Week 1 | 0.03 (0.01) | 0.00 (0.01)
  Change at Week 2 | 0.03 (0.01) | 0.00 (0.01)
  Change at Week 3 | 0.08 (0.03) | 0.00 (0.03)
  Change at Week 4 | 0.05 (0.02) | 0.00 (0.02)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.145, Mixed Models Analysis; Difference in LS mean = 0.03, 95% CI 2-sided [-0.01 to 0.06], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.148, Mixed Models Analysis; Difference in LS mean = 0.03, 95% CI 2-sided [-0.01 to 0.07], Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.082, Mixed Models Analysis; Difference in LS mean = 0.07, 95% CI 2-sided [-0.01 to 0.15], Standard Error of Mean 0.04
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.070, Mixed Models Analysis; Difference in LS mean = 0.04, 95% CI 2-sided [-0.00 to 0.09], Standard Error of Mean 0.02

ADVERSE EVENTS:
Time Frame: Screening (2 Weeks prior to Day 1) up to maximum of 5 Weeks after administration of the final dose of study medication (maximum up to 11 weeks)
Description: Same event may appear as both AE and SAE. An event may be categorized as serious in 1 participant and non-serious in other, or participant may experience both SAE and non-SAE.
Arm/Group | Ziprasidone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/85
Serious Adverse Events (participants affected / at risk) | 3/86 | 0/85
Other Adverse Events (participants affected / at risk) | 65/86 | 35/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=86) | Placebo (N=85)
Chest pain (General disorders) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=86) | Placebo (N=85)
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 12 | 5
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 9 | 3
Fatigue (General disorders) | 19 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 10 | 0
Increased appetite (Metabolism and nutrition disorders) | 3 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Akathisia (Nervous system disorders) | 5 | 0
Dizziness (Nervous system disorders) | 6 | 2
Headache (Nervous system disorders) | 9 | 8
Hypersomnia (Nervous system disorders) | 2 | 0
Sedation (Nervous system disorders) | 8 | 3
Somnolence (Nervous system disorders) | 27 | 7
Speech disorder (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 0 | 4
Anxiety (Psychiatric disorders) | 3 | 0
Initial insomnia (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Irritability (Psychiatric disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT02075047/Prot_001.pdf
  • Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT02075047/SAP_000.pdf